CLINICAL TRIAL: NCT00136500
Title: Clinical Research in Amyotrophic Lateral Sclerosis
Brief Title: Clinical Research in ALS Study
Acronym: CRiALS
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: ALS Association (Other); ALS Recovery Fund (Unknown)
Responsible Party: Principal Investigator, Michael Benatar, Professor, University of Miami
Other Study IDs: 20101021
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: genetics; biomarkers; pre-symptomatic; natural history
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, blood, urine, CSF, skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Individuals affected with ALS: This population be sporadic or familial ALS.
- Unaffected individuals from families in which the genetic cause of ALS is known: This population includes pre-symptomatic individuals at genetic risk for ALS or a related neurodegenerative disorder (i.e., FTD).
- Individuals affected with an ALS-related neurodegenerative disease: This would include FTD, MSP, IBMPFD, etc.
- Healthy controls

SUMMARY:
CRiALS is an umbrella protocol through which people are recruited to participate in a range of research studies being conducted by the ALS Research Collaboration (ARC).

DETAILED DESCRIPTION:
Research goals include elucidation of the complex relationship between ALS and related neurodegenerative disorders, development of both wet and dry biomarkers of disease, and delineation of the full course of the natural history of disease from the early pre-symptomatic stages through established and even late-stage disease. These goals are accomplished through the recruitment and evaluation of patients with ALS and related diseases, family members (including people at genetic risk for ALS, but who are not yet affected), and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Member of at least one of the following categories:

   1. Individuals affected with ALS or a related neurodegenerative disease (sporadic or familial)
   2. Unaffected individuals from fALS pedigrees, including pre-symptomatic individuals at genetic risk for ALS or individuals from pedigrees of ALS related diseases.
   3. Healthy controls
3. Able and willing to comply with relevant procedures.

Exclusion Criteria:

1. Subject has a condition or is in a situation which, in the PI's opinion, could confound the study finding or may interfere significantly with the individual's participation and compliance with the study protocol -- including but not limited to neurological, psychological and/or medical conditions (e.g., multiple sclerosis, neuropathy, myelopathy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The CRiALS research program aims to recruit three types of participants:
  * Individuals affected with ALS or a related neurodegenerative disease
  * Unaffected individuals from pedigrees in which the genetic cause of ALS is known
  * Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2005-02; Primary Completion 2037-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Annually
  Since this is an umbrella/gateway protocol through which individuals are recruited to participate in a range of studies, outcome is assessed in terms of recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Benatar, MD, PhD., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ALS Research Collaboration — http://als-research.org/